CLINICAL TRIAL: NCT07379385
Title: The Effect of Weekly Set Volume of Resistance Training on Strength and Hypertrophy
Brief Title: Effects of Weekly Set Volume on Muscle Adaptation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Andreo Fernando Aguiar, Principal Investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Weekly set volume study
Record Dates: First submitted 2026-01-07; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Muscle Performance; Resistance Training
Keywords: Resistance exercise; Weekly set volume; Training volume; Muscle hypertrophy; Muscle strength; Aging
MeSH Terms: interventions — Hospitals, Low-Volume; Hospitals, High-Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Volume (LV) (Experimental): Participants will be performed 6 sets/week
  Interventions: Other: Low volume (LV)
- Moderate Volume (MV) (Experimental): Participants will be performed 18 sets/week
  Interventions: Other: Moderate Volume (MV)
- High Volume (HV) (Experimental): Participants will be performed 30 sets/week
  Interventions: Other: High Volume (HV)

INTERVENTIONS:
Other: Low volume (LV) — Participants will be performed 6 sets/week during 10 weeks
  Arms: Low Volume (LV)
Other: Moderate Volume (MV) — Participants will be performed 18 sets/week during 10 weeks
  Arms: Moderate Volume (MV)
Other: High Volume (HV) — Participants will be performed 30 sets/week during 10 weeks
  Arms: High Volume (HV)

SUMMARY:
The progressive loss of strength and muscle mass is a natural aging process, with direct implications for functional capacity. Resistance training (RT) is considered the main intervention to counteract this decline. Although the RT guidelines are well established, the ideal weekly set volume to maximize strength and hypertrophy gains in older adults remains unknown. The purpose of this study is to investigate the effects of different volumes of weekly sets of RT on muscle strength and hypertrophy in older adults

DETAILED DESCRIPTION:
BACKGROUND: The progressive loss of strength and muscle mass is a natural process of aging, with direct implications for functional capacity. Resistance training (RT) is considered the main intervention to counteract this decline. Although RT guidelines are well established, the ideal weekly volume of sets to maximize strength and hypertrophy gains in older adults remains unknown. PURPOSE: To investigate the effects of different weekly RT volumes on lower limb muscle strength and hypertrophy (quadriceps femoris) in older adults. METHODS: Fifty-seven older adults of both sexes will be matched for maximum dynamic strength (one repetition maximum - 1RM) and randomly divided into 03 groups: [Low Volume (LV = 6 sets/week, n = 19), Moderate Volume (MV = 18 sets/week, n = 19) and High Volume (LV = 30 sets/week, n = 18)]. All participants will undergo a 10-week resistance training protocol (3x/week), consisting of 8 exercises: bench press, leg press, seated row, leg extension, bicep curl, leg curl, triceps pulley, and seated calf raise. Only the leg extension and leg press exercises will be performed with different volumes of sets (VB = 1 set/exercise; VM = 3 sets/exercise; VA = 5 sets/exercise). The number of repetitions per set will be 8-12, and the training load will be adjusted every two weeks based on the maximum number of repetitions performed in the last training session. The following dependent variables will be analyzed before and after the training program: (1) maximum dynamic strength (1RM) and (2) maximum voluntary isometric contraction (MVIC) in the leg extension exercise, (3) muscle hypertrophy (thickness) of the quadriceps muscle and rectus femorisusing ultrasound images, and (4) rating of perceived exertion (RPE) and (5) affective responses (pleasure and displeasure) after training sessions. Data will be tested for normality and homogeneity using the Shapiro-Wilk's and Levene's tests, respectively. Changes over time and between groups will be analyzed with two-way repeated measures ANOVA tests. Violation of sphericity was corrected using the Greenhouse-Geisser method. When significant differences will be confirmed with the ANOVA, multiple comparison testing will be performed using the Bonferroni post hoc correction to identify these differences. Values will be expressed as mean (standard deviation and 95% confidence interval). The significance level was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 80 years

Exclusion Criteria:

* not having used any medication or substance that affects or improves muscle function for at least 3 months prior to the study,
* having any physical or physiological limitation that may affect the ability to perform the tests and physical training,
* not being able to understand the informed consent form and study procedures.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Maximum dynamic strength (1RM) | baseline and after 10 weeks of intervention
  The one-repetition maximum test will be performed on a bilateral leg extension machine. Briefly, participants will undergo 3 test attempts, interspersed with 5-minute intervals. Loads of 10-15% will be added after each attempt in order to reach the 1RM load within the 3 trials. Participants will be verbally encouraged during each attempt.
Maximum voluntary isometric contraction (MVIC) | baseline and after 10 weeks of intervention
  The MVIC test for the leg extension exercise (bilateral) will be performed using an isometric dynamometer (CEFISE Biotechnology, São Carlos, Brazil). Briefly, participants will perform three MVICs at 120º of knee flexion (180º = full extension) lasting 5 s, interspersed with 5 s of rest. Participants will be instructed and verbally encouraged to exert maximum force during all attempts. The highest value obtained for peak and mean torque of the three MVICs will be used for the analysis.
Muscle hypertrophy (thickness) | baseline and after 10 weeks of intervention
  Muscle hypertrophy (thickness) of the quadriceps and rectus femoris muscles will be assessed using ultrasound images obtained at 3 anatomical points (30, 50, and 60% of the distance between the greater trochanter of the femur and the knee joint line). Muscle thickness will be analyzed using the image analysis program (ImageJ®).

SECONDARY OUTCOMES:
Rating of perceive exterion (RPE) | Immediately after completion of each set of exercise
  Rating of perceived exertion (RPE) will be recorded immediately after completion of each set using the OMNI-RES scale. The participants will be instructed to report the perceived exertion value by indicating a number on the OMNI-RES scale (0 for ''no effort'' and 10 for ''maximal effort'') that best represented their momentary exertion.
Affective responses (pleasure and displeasure) | Immediately after each exercise during training sessions
  The affective response will be assessed using an 11-point affectivity scale, ranging from +5 to -5, with a score of zero considered neutral, positive numbers (+1 to +5) representing feelings of pleasure, and negative numbers (-1 to -5) representing feelings of displeasure.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern University of Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robertson RJ, Goss FL, Rutkowski J, Lenz B, Dixon C, Timmer J, Frazee K, Dube J, Andreacci J. Concurrent validation of the OMNI perceived exertion scale for resistance exercise. Med Sci Sports Exerc. 2003 Feb;35(2):333-41. doi: 10.1249/01.MSS.0000048831.15016.2A. PMID 12569225